CLINICAL TRIAL: NCT07046221
Title: Tislelizumab Combined With Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma Followed by CRT or Surgery: A Prospective, Open-label, Multicenter Clinical Study
Brief Title: Tislelizumab Combined With Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma Followed by CRT or Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-01
Record Dates: First submitted 2025-06-15; First posted 2025-07-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; Albumin-Bound Paclitaxel; Cisplatin; Surgical Procedures, Operative; Radiation; nedaplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT+Tislelizumab (Experimental): RT：50.5Gy/28f albumin-bound paclitaxel：125mg/m2，d1，d8，q3w，2cycles cis-platinum：75mg/m2，d1，q3w，2cycles/carboplatin：AUC=5，d1，q3w，2 cycles/Nedaplatin：80-100mg/m2，d1，q3w，2 cycles Tislelizumab: 200mg，d1，q3w，1years
  Interventions: Drug: Tislelizumab; Drug: Albumin-Bound Paclitaxel; Drug: cis-platinum; Radiation: Radiation; Drug: Nedaplatin; Drug: Carboplatin
- surgery+Tislelizumab (Experimental): Radical resection of esophageal cancer Tislelizumab: 200mg，d1，q3w，1years
  Interventions: Drug: Tislelizumab; Procedure: Surgery

INTERVENTIONS:
Drug: Tislelizumab — 200mg，d1，q3w，1years
Drug: Albumin-Bound Paclitaxel — 125mg/m2，d1，d8，q3w，2cycles
  Arms: CRT+Tislelizumab
Drug: cis-platinum — 75mg/m2，d1，q3w，2cycles
  Arms: CRT+Tislelizumab
Procedure: Surgery — Radical resection of esophageal cancer
  Arms: surgery+Tislelizumab
Radiation: Radiation — 50.5Gy/28f
  Arms: CRT+Tislelizumab
Drug: Nedaplatin — 80-100mg/m2，d1，q3w，2cycles
  Arms: CRT+Tislelizumab
Drug: Carboplatin — AUC=5，d1，q3w，2cycles
  Arms: CRT+Tislelizumab

SUMMARY:
To explore the non-inferiority of the 2y-OS rate of tislelizumab combined with chemotherapy after sequential CRT in the treatment of resectable esophageal squamous cell carcinoma compared with the surgical group

ELIGIBILITY:
Inclusion Criteria:

* The subjects were included in this study and signed the informed consent form.
* Male or female patients aged between 18 and 75 years old;
* Patients diagnosed with esophageal squamous cell carcinoma by histopathology;
* According to the 8th edition of the AJCC Esophageal cancer TNM staging system, it is located in cT2N+ or cT3-4aNanyM0 (confirmed by enhanced CT/MRI of the chest and abdomen), and the lesion is located in the thoracic segment.
* ECOG score: 0-1.
* The main organs function normally, that is, they meet the following standards:

  1. Blood routine (no blood transfusion was performed within 14 days before treatment, no granulocyte colony-stimulating factor [G-CSF] was used, and no other drugs were used for correction);

     The absolute neutrophil count (ANC) was ≥1.5×109/L;

     Hemoglobin (HB) ≥9.0 g/dL;

     Platelet count (PLT) ≥100×109/L;
  2. Blood biochemistry

Creatinine clearance rate ≥60 mL/min;

Total bilirubin (TBIL) ≤ 1.5×ULN;

Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤2.5×ULN;

* The expected survival period is ≥3 months;
* Female subjects with reproductive capacity and male subjects whose partners are of childbearing age need to adopt a medically approved contraceptive measure during the study treatment period and for at least 3 months after the last treatment

Exclusion Criteria:

* There are clinically uncontrolled pleural effusions, pericardial effusions or ascites that require repeated drainage or medical intervention (within 2 weeks before randomization);
* It is known that there is intolerance or resistance to the chemotherapy specified in the trial protocol;
* Have received any other ESCC anti-tumor treatments (e.g., targeted treatments for PD-1, PD-L1, PD-L2, or other tumor immunotherapy, radiotherapy, targeted therapy, ablation, or other systemic or local anti-tumor treatments);
* Patients with active autoimmune diseases or a history of autoimmune diseases that may recur, or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Have a history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including pulmonary fibrosis, acute lung diseases, etc.
* Before enrollment, there was a severe chronic or active infection (including tuberculosis infection, etc.) that required systemic antibacterial, antifungal or antiviral treatment;
* A known history of HIV infection;
* Having suffered from other malignant tumors within the past five years (excluding cured basal cell carcinoma of the skin, carcinoma in situ of the breast and carcinoma in situ of the cervix);
* Have received live vaccines within 28 days before enrollment;
* Participated in other therapeutic clinical trials within 4 weeks;
* Those that the researchers consider unsuitable for inclusion.
* Distant metastasis exists (except for supraclavicular lymph nodes).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate of 2 years | 2 years
  The proportion of patients who were still alive from the start of randomization (or the start of treatment in a single-arm trial) to 2 years

SECONDARY OUTCOMES:
objective response rate | every 2 weeks until 3 years
  According to the recognized response evaluation criteria (such as recist Version 1.1 for Solid tumors), the proportion of patients whose tumor volume reduction reaches the pre-specified value and can maintain the minimum time limit requirements